CLINICAL TRIAL: NCT04791163
Title: AK Socket Evaluation : Sub-ischial vs Ischial Containment. Multi-center Randomised Crossover Study
Brief Title: Above-knee Socket Evaluation : Sub-ischial vs Ischial Containment
Acronym: P20-EMBSUBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteor Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A03303-36
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-ischial socket (Experimental): Start using the sub-ischial socket for four weeks and be tested with this socket.
  Interventions: Device: Socket evaluation
- Ischial containment socket (Active Comparator): Start using the ischial containment socket for four weeks and be tested with this socket.
  Interventions: Device: Socket evaluation

INTERVENTIONS:
Device: Socket evaluation — The subject will wear the socket for 4 weeks, and then reply questionnaires and achieve a 2-minute walking test

SUMMARY:
Socket is key to provide comfort and function to lower limb amputees. A new socket, the sub-ischial socket, will be compared to "traditional" ischial containment sockets, based on comfort self-evaluation, and locomotor capacities.

DETAILED DESCRIPTION:
Subjects wearing ischail containment sockets will be proposed to enter the research. They will be provided and fitted with a sub-ischial socket. Randomly, they will use one or the other socket for four weeks, then be tested : finctional test and questionnaires. After this testing session, they will use the other socket, and be re-tested accordingly.

ELIGIBILITY:
Inclusion Criteria:

* can give informed consent
* aged 18 or more
* above-knee amputee, wearing a definitive ischial containment socket
* stump longer than 16cm
* wearing a liner, whatever the suspension system
* able to walk (d4600, d4601, d4602, d4608 accordinf to IFC)
* unilaterla or bilateral amputee
* able to done the socket standing
* whatever the etiology

Exclusion Criteria:

* protected person
* pregnant woman or nursing mother
* subject having comorbidities heavily impacting feeling or socket donning
* allergic to silicon
* suffering from big volume variations in a same day
* infecté stump (may lead to lymphatic problems)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Comfort evaluation | 1 minute
  Socket Comfort Score (SCS)

SECONDARY OUTCOMES:
Comfort evaluation in various situations | 1 minute
  Same question for four detailed situations
Locomotor capability | 5 minutes
  PLUS-M questionnaire and 2-minute walking test

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Les Capucins, Angers
  - UGECAM La Tour de Gassies, Bruges
  - Clinique du Cabirol, Colomiers
  - Hôpital Léon Bérard, Hyères
  - UGECAM - IRR Nancy, Nancy
  - Institution Nationale des Invalides, Paris
  - Centre Mutualiste de Kerpape, Ploemeur
  - UGECAM La Tourmaline, Saint-Herblain
  - CHBA Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No